CLINICAL TRIAL: NCT03593616
Title: Auditing of Poor Visual Outcomes After Un-eventual Cataract Surgery: a Prospective Cohort Study
Brief Title: Auditing of Poor Visual Outcomes After Un-eventual Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Abd Elkafy, Principal investigator, Assiut University
Other Study IDs: UECS
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lens Phacoemulsification Group: insertion of intra-ocular lens
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — insertion of intra-ocular lens after emulsification of catractous lens

SUMMARY:
Globally, cataract is the major cause of blindness accounting for 51% of total blindness and there are regional variations in it. Today, cataract surgery is a highly successful and cost-effective procedure, which enhances both the vision and quality of life of patients.

Visual acuity alone should not be used as a criterion for planning cataract surgery, since visual acuity and function do not necessarily correlate. Therefore, there is a need to review our criteria for management.

Based on recent studies, at least 90% of the patients undergoing cataract surgery obtain a postoperative visual acuity of 6/12 or better in the absence of coexisting ocular pathology.

A number of previous studies have looked at the effect of risk factors on visual outcomes following cataract surgery. Risk factors commonly associated with worse visual outcomes include: age-related macular degeneration, diabetic retinopathy, corneal opacity/pathology, older age, female sex, previous vitrectomy, previous retinal detachment surgery, alpha-blockers, complex surgery, intraoperative complications and refractive surprise.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any type of cataract.

Exclusion Criteria:

* Patients with diabetic retinopathy.
* Patients with previous ocular surgeries or pathologies.
* Patients with pre-operative visual acuity (no perception of light)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients for cataract surgery received a comprehensive ophthalmic examination. The standard pre-operative examination included a detailed history, measurements of presenting visual acuity
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The visual acuity of patients after cataract surgery | 4 weeks
  measured by snellen's chart

IPD SHARING:
Plan to Share IPD: Undecided